CLINICAL TRIAL: NCT06890078
Title: Optimisation du Diagnostic de Pneumocystose Chez Les Patients Immunodéprimés
Brief Title: Optimizing the Diagnosis of Pneumocystis in Immunocompromised Patients
Acronym: OPTIJIROVEC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231319
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pneumocystis; Immunocompromised Patients
Keywords: immunocompromised patients; pneumocystis
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mouthwash, throat swab, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with suspicion of pneumocystis
  Interventions: Other: Biological sampling

INTERVENTIONS:
Other: Biological sampling — Mouthwash, nasopharyngeal swab, blood sampling

SUMMARY:
Evaluate new diagnostic methods using qPCR on non-invasive samples, compared with reference techniques for the positive diagnosis of pneumocystis (PcP) in immunocompromised patients

ELIGIBILITY:
Inclusion Criteria:

* adult patients with suspected pneumocystis
* with an indication for bronchial fibroscopy for BAL or induced sputum
* no opposition to the research from the adult patient or his or her next of kin research for patients unable to express their non-opposition

Exclusion Criteria:

* Pneumocystis treated for more than 72 hours
* pregnancy/breast-feeding
* adult patients deprived of liberty, protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected pneumocystis
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Pearson correlation coefficient | At inclusion
  Pearson correlation coefficient between the fungal load obtained by PCR on nasopharyngeal swabs nasopharyngeal swab and buccal lavage and that obtained by reference samples (induced sputum or BAL) in patients with confirmed PcP.

SECONDARY OUTCOMES:
Fungal load by qPCR | At inclusion
  Quantitative fungal load results obtained by qPCR on nasopharyngeal swab, mouthwash, induced sputum, BAL
Fungal load by serum PCR | At inclusion
  Quantitative fungal load results obtained by serum PCR
Beta D glucan blood levels | At inclusion

IPD SHARING:
Plan to Share IPD: Undecided